CLINICAL TRIAL: NCT04473287
Title: The Effect of Reflexology Applied to Patients Undergoing Coronary Artery Bypass Graft Surgery on Pain, Anxiety, Fatigue and Sleep: A Randomized Controlled Study
Brief Title: The Effect of Reflexology After Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, PhD, Asst Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-10/35
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: reflexology, pain, anxiety, fatigue, sleep
MeSH Terms: conditions — Pain; Anxiety Disorders; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Reflexology was applied to the intervention group during the procedure for 45 minutes.
  Interventions: Other: reflexology practice
- control group (No Intervention): Reflexology was not applied to the control group during the procedure. The control group received standard care and treatment.

INTERVENTIONS:
Other: reflexology practice — Reflexology is a reliable and holistic complementary and alternative treatment method that means that the body's specific glands, organs and regions are stimulated by applying a special pressure with the fingers on the hands, feet and ears. When the literature is analyzed, it has been determined that reflexology is applied effectively before, during and after surgery, including different surgical procedures, and it is emphasized that one of the most important areas is patients who underwent Coronary Artery Bypass Graft (CABG) surgery. In this study, it is thought that reflexology application to patients undergoing CABG surgery on nursing care will contribute to the nursing literature by examining the effect of reflexology on pain, anxiety, fatigue, sleep and physiological parameters.
  Arms: intervention group

SUMMARY:
Coronary artery bypass graft (CABG) surgery is a treatment method that increases survival rate in the treatment of coronary artery disease (CAD). CABG surgery can create anxiety, fear, pain, fatigue, sleep disorders and physiological dysfunctions in patients. Nurses responsible for the care and treatment of patients use pharmacological and non-pharmacological methods to alleviate the problems that arise. In this context, reflexology within complementary and alternative therapy (CAM) can be applied. In this study, it is aimed to evaluate the effect of reflexology applied to patients undergoing coronary artery bypass graft surgery on pain, anxiety, fatigue, sleep and physiological parameters.

DETAILED DESCRIPTION:
In the literature, there are a limited number of studies on the effect of reflexology applied on patients undergoing CABG surgery on anxiety and physiological parameters. In addition, no studies on the effect of reflexology on sleep on patients undergoing CABG surgery have been encountered. Anxiety, stress, pain, fatigue, sleep disorders and permanent symptoms may occur in individuals after cardiovascular surgery. It has been determined that with the deterioration in the body system functions and the resulting psychological problems, the blood pressure, heart rhythm and the number of breaths in the individual, respiratory and coughing difficulties due to pain inactivity, body temperature changes, muscle tension, fatigue and even death can occur. With the application of reflexology, the work of the body systems is regulated by providing homeostasis, physiological and psychological relaxation and relaxation are felt with the energy flow that occurs in the body, and toxins are removed from the body. In this study, it is thought that reflexology application to patients undergoing CABG surgery on nursing care will contribute to the nursing literature by examining the effect of reflexology on pain, anxiety, fatigue, sleep and physiological parameters. The population of the study will be the patients who underwent CABG surgery in the Cardiovascular Intensive Care Unit and Cardiovascular Surgery Clinic of Uludağ University Health Practice and Research Center Hospital. The sample will be composed of patients undergoing CABG surgery in Uludag University Health Practice and Research Center Hospital Cardiovascular Surgery Department Cardiovascular Intensive Care Unit and Cardiovascular Surgery Clinic that meet the inclusion criteria. Data will be collected using Personal Information Form, Physiological Parameters Control Form, Visual Analogue Scale, State Anxiety Scale, Richard's Campbell Sleep Scale. The data obtained from the research will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Number, percentage, average and standard deviation will be used as descriptive statistical methods in the evaluation of the data. The t-test will be used to compare quantitative continuous data between two independent groups. Differences between repeated measurements will be analyzed by repeated measurements ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having undergone CABG surgery for the first time
* CABG has not been operated in an emergency
* Lack of reflexology history
* Not taking inotropic drugs At least 4 hours have passed since the application of the last analgesic drug
* Mental insufficiency and no vision, hearing impairment
* Place, time and person orientation
* Psychological treatment and drug use for this purpose
* Participants agree to participate in the research

Exclusion Criteria:

* Decreased level of consciousness
* Valve repair or replacement during CABG surgery Need for intraaortic balloon and pacemaker
* Drainage over 200 ml per hour
* Having a history of chronic pain
* Being addicted to alcohol and drugs
* Bone fractures, sensory disorders, skin infections, skin ulcers in the feet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change on pain intensity as measured by Visual Analog Scale | ''just before procedure'' and ''30 minutes after procedure''
  The average score change on pain intensity as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure pain intensity. The scale is a measuring tool with length of 0-10 cm. High scores on the scale indicate that pain intensity is high.
Change on fatigue intensity as measured by Visual Analog Scale | ''just before procedure'' and ''30 minutes after procedure''
  The average score change on fatigue intensity as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure fatigue intensity. The scale is a measuring tool with length of 0-10 cm. High scores on the scale indicate that fatigue intensity is high.

SECONDARY OUTCOMES:
Score change on anxiety level as measured by State-Trait Anxiety Inventory | ''just before procedure'' and ''30 minutes after procedure''
  The average score change on anxiety level as measured by State-Trait Anxiety Inventory. This scale in used to measure anxiety. The scores on the scale ranges from 20 to 80. The high scores on the scale indicate that anxiety is high.
Score change on sleep quality as measured by Richard's Campbell Sleep Scale | ''just before procedure'' and ''30 minutes after procedure''
  The average score change on sleep quality as measured by Richard's Campbell Sleep Scale. This scale in used to measure sleep quality. The scores on the scale ranges from 0 to 100. The high scores on the scale indicate that sleep quality is high.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, RN, PhD, Principal Investigator — Sağlık Bilimleri Üniversitesi, Turkey
Locations (1):
- Sağlık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bagheri-Nesami M, Shorofi SA, Zargar N, Sohrabi M, Gholipour-Baradari A, Khalilian A. The effects of foot reflexology massage on anxiety in patients following coronary artery bypass graft surgery: a randomized controlled trial. Complement Ther Clin Pract. 2014 Feb;20(1):42-7. doi: 10.1016/j.ctcp.2013.10.006. Epub 2013 Oct 25. PMID 24439644
- [Result] Abbaszadeh Y, Allahbakhshian A, Seyyedrasooli A, Sarbakhsh P, Goljarian S, Safaei N. Effects of foot reflexology on anxiety and physiological parameters in patients undergoing coronary artery bypass graft surgery: A clinical trial. Complement Ther Clin Pract. 2018 May;31:220-228. doi: 10.1016/j.ctcp.2018.02.018. Epub 2018 Mar 3. PMID 29705459
- [Result] Tully PJ, Bennetts JS, Baker RA, McGavigan AD, Turnbull DA, Winefield HR. Anxiety, depression, and stress as risk factors for atrial fibrillation after cardiac surgery. Heart Lung. 2011 Jan-Feb;40(1):4-11. doi: 10.1016/j.hrtlng.2009.12.010. Epub 2010 May 8. PMID 20561864
- See also: The Effects of Foot Reflexology Massage on Pain and Fatigue of Patients After Coronary Artery Bypass Graft — http://jmums.mazums.ac.ir/files/site1/user_files_0d0bf0/bmahmadi-A-10-1768-57-5d57eec.pdf
- See also: An Alternative Method for Labor Pain: Foot Reflexology — http://hacettepehemsirelikdergisi.org/pdf/pdf_HHD_230.pdf